CLINICAL TRIAL: NCT03252262
Title: Power V360 - Promoting Optimal Wellness Among Elders Through Vitalize 360
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P 30 AG048785
Record Dates: First submitted 2017-04-12; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-04

CONDITIONS: Health, Subjective

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jack Satter House (Active Comparator): Residents of Jack Satter House who participated in the Vitalize 360 Program.
  Interventions: Other: Vitalize 360
- Center Communities of Brookline (Active Comparator): Residents of Center Communities of Brookline who participated in the Vitalize 360 Program.
  Interventions: Other: Vitalize 360
- Simon C. Fireman (Active Comparator): Residents of Simon C. Fireman who participated in the Vitalize 360 Program
  Interventions: Other: Vitalize 360

INTERVENTIONS:
Other: Vitalize 360 — A comprehensive geriatric assessment system and wellness coaching program.

SUMMARY:
The primary purpose of this project was to implement Vitalize 360, a comprehensive assessment system and wellness coaching program for vulnerable, low income, community dwelling older adults, and to determine if this program is effective in promoting and sustaining self-management skills to increase well-being and functional health among this group. Designed specifically for community-dwelling older adults, Vitalize 360 provides a unique opportunity to guide elders in selecting personal goals that align with their assessment results and develop an action plan for goal achievement. This strategy holds potential as an effective mechanism to empower elders to implement behaviors that promote healthy aging.

DETAILED DESCRIPTION:
The purpose of this project was to determine if Vitalize 360, a comprehensive assessment system and wellness coaching program was effective in promoting and sustaining increased physical activity and improved mood, health status and quality of life. A repeated measures, secondary analysis design was the selected approach Data from 161 participants were used to test the hypotheses. After one year, the sample had improvement with increased socialization while physical activity level fluctuated over time suggestive of a seasonality effect. Paired t-tests and repeated measures analysis revealed no statistically significant improvement in physical activity level, mood, health status or quality of life. Vitalize 360 provides a unique opportunity to guide elders in selecting personal goals that align with their assessment results and develop an action plan for goal achievement. When used among vulnerable and frail elders, some modifications are needed to provide sustained, favorable outcomes.

ELIGIBILITY:
Inclusion Criteria:

Age 60 years and over, residing in subsidized housing sites operated by Hebrew SeniorLife and participating in Vitalize 360 program

Exclusion Criteria:

younger than 60 years, not participating in Vitalize 360 program and not a permanent resident of housing sites.

Min Age: 60 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | 18 months
  number of hours engaged in physical activity over the past 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth P Howard, PhD, Principal Investigator — Hebrew Rehabilitation Center

IPD SHARING:
Plan to Share IPD: Yes
Contact PI to obtain approval for use of COLLAGE/interRAI data